CLINICAL TRIAL: NCT03626610
Title: 'Pre-EMPT' - An Interventional Study to Assess the Effects of Pre-emptive Exercise , or 'Prehabilitation', in Patients Undergoing Peri-operative Treatment for Adenocarcinoma of the Oesophagus and Gastro-oesophageal Junction
Brief Title: Prehabilitation of Patients With oEsophageal Malignancy Undergoing Peri-operative Treatment
Acronym: Pre-EMPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRAS 204711 Pre-EMPT PROTOCOL
Record Dates: First submitted 2018-07-24; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Oesophageal Adenocarcinoma; Chemotherapy Effect; Surgery
Keywords: Prehabilitation; Exercise; Cancer; Neo-adjuvant chemotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Motor Activity; Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort-controlled
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Participants will be given a monitored exercise program during their treatment starting before chemotherapy
  Interventions: Behavioral: Exercise prehabilitation during chemotherapy before surgery
- Non-interventional (No Intervention): Patients will have standard care.

INTERVENTIONS:
Behavioral: Exercise prehabilitation during chemotherapy before surgery — Monitored exercise training in patients with a new diagnosis of oesophageal adenocarcinoma
  Arms: Interventional

SUMMARY:
'Pre-EMPT' - A cohort-controlled, interventional study to assess the effects of a pre-emptive exercise programme, or 'prehabilitation', in patients undergoing peri-operative chemotherapy for adenocarcinoma of the lower oesophagus and gastro-oesophageal junction.

DETAILED DESCRIPTION:
Oesophageal cancer has the fastest rising incidence of any solid tumour in the western world with the UK, and London, having particularly high rates of the disease.

Those patients being considered for "cure" will benefit from pre-operative/neo-adjuvant chemotherapy (NAC), which is known to have a deleterious effect on fitness and is associated with increased post-operative morbidity. Post-operative morbidity is also associated with reduced survival. Reduction in fitness is compounded by major surgery and significantly reduces the numbers of patients who commence or complete the standard treatment of post-operative chemotherapy to around 40%.

Chemotherapy and surgery for oesophageal cancer both represent significant physiological insults that may have detrimental effects on physical activity and outcomes after surgery. Cardiopulmonary exercise (CPEX) testing has been effectively used in numerous tumour groups to predict outcome after surgery, although its role in oesophageal cancer patients remains uncertain owing to conflicting data from institutional series. Advanced exercise programmes, sometimes termed 'prehabilitation', directed by experienced multidisciplinary teams are increasingly being used to mitigate the secondary effects of cancer treatment.

'Prehabilitation' has been shown to reduce postoperative morbidity and mortality in thoracic patients undergoing elective high-risk surgery. In addition, results of studies examining physical exercise and cancer recurrence/survival which effect immune system function in cancer survivors suggest that physical exercise training may improve a number of immune system parameters that may be important in cancer defence.

The investigators believe that optimising patient fitness through a structured and expert-devised exercise programme of 'prehabilitation' during neo-adjuvant chemotherapy and prior to surgery will mitigate the effects of chemotherapy and improve patient outcomes after surgery.

The investigators intend to assess the feasibility of a 'prehabilitation' programme and quantify the resultant effects primarily using CPEX testing. In addition, changes in hospital 'length of stay' will be documented with a number of additional parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed with operable oesophageal and gastro-oesophageal adenocarcinoma and scheduled to undergo standard neo-adjuvant chemotherapy and oesophago-gastric surgery as recommended by the Multidisciplinary Meeting decision.
2. 18+
3. </=79 (patients above this age may be included in studies after the feasibility study has been completed)
4. Participants must be able to understand and independently consent to participation in the study.
5. Participants must be able to understand and complete the questionnaires.
6. Participants must be willing to undergo all the standard assessments and interventions included in this study - CPEX testing, blood sampling, questionnaires and exercise intervention where appropriate.
7. Participants must be willing to wear the Fibit monitoring device and agree with its use
8. Participants must be ASA 1-3 and fit for surgical resection
9. Patients should have a Body Mass Index (BMI) equal to or above 18.5 with less than 10% self-reported unintentional weight loss at diagnosis.

Exclusion Criteria:

Participants will be excluded if they:

1. Are not considered medically fit for surgery at diagnosis, as decided by the Multidisciplinary team
2. Will undergo primary or palliative chemotherapy
3. Are recommended to have chemoradiotherapy
4. Are under 18 years old
5. Are over 79 years old
6. Are unable to undergo CPEX testing
7. Do not wish to take part in selected aspects of the study
8. Cannot or do not wish to attend the CHHP for assessment and/or advice on exercise
9. Cannot understand and give informed consent to the study
10. Cannot understand and complete the questionnaires
11. Do not wish to wear a Fitbit monitoring device
12. ASA 4+
13. Patients with BMI of less than 18.5 with self-reported unintentional weight loss of 10% or more at diagnosis.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary fitness | Baseline to 5 months
  Cardiopulmonary exercise test on bicycle ergometer

SECONDARY OUTCOMES:
Post-operative complications | Date of surgery to date of discharge, up to 45 days post-surgery
  Clavien-Dindo; ECCG- Esophageal Complications Consensus Group
Post-operative length of hospital stay | Date of surgery to date of discharge, up to 45 days post-surgery
  Number of in-hospital days from date of surgery
Lean body mass | Baseline to 5 months
  Computerised tomography assessment of lean body mass
Daily activity levels | Baseline to 5 months
  Steps per day measured by Fitbit
Sleep quality assessment | Baseline to 5 months
  Sleep data from Fitbit
Change in Health-related Quality of Life: Oesophageal cancer-specific questionnaire | Baseline to 12 months post-surgery
  EORTC QLQ-OES18
Change in Health-related Quality of Life: Cancer questionniare | Baseline to 12 months post-surgery
  EORTC QLQ-C30
Change in Well-being | Baseline to 12 months post-surgery
  SWEMWEBS questionnaire
Disease recurrence | Date of surgery to date of recurrence, up to 12 months post-surgery
  Pathological or radiological confirmation of recurrent disease
Post-operative mortality | Date of surgery to date of death, up to 12 months post-surgery
  In-patient, 30-day, 90-day, 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MBChBMDFRCS, Principal Investigator — Consultant Surgeon
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zylstra J, Whyte GP, Beckmann K, Pate J, Santaolalla A, Gervais-Andre L, Russell B, Maisey N, Waters J, Tham G, Lagergren J, Green M, Kelly M, Baker C, Van Hemelrijck M, Goh V, Gossage J, Browning M, Davies A. Exercise prehabilitation during neoadjuvant chemotherapy may enhance tumour regression in oesophageal cancer: results from a prospective non-randomised trial. Br J Sports Med. 2022 Apr;56(7):402-409. doi: 10.1136/bjsports-2021-104243. Epub 2022 Feb 1. PMID 35105604